CLINICAL TRIAL: NCT00831571
Title: Prospective Analysis of Hypersensitivity Reactions to Oxaliplatin
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 08-140; SANOFI OX-07-008
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Small Bowel Cancer; Pancreatic Cancer
Keywords: oxaliplatin; hypersensitivity
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- All Participants: Patients receiving Oxaliplatin
- Desensitization: Patients that have experienced a moderate to severe hypersensitivity reaction to oxaliplatin

SUMMARY:
This research study will examine how often hypersensitivity, or allergic reactions, occur in patients receiving the chemotherapy medication oxaliplatin. Hypersensitivity reactions can vary from a transient skin rash and fever to more severe symptoms such as shortness of breath, chest tightness, and a more severe allergic reaction that can affect blood pressure called anaphylaxis. We will be examining how often hypersensitivity reactions occur and how severe the reactions are when they occur. We will also examine whether there are factors that place people at risk for developing hypersensitivity reactions to oxaliplatin. In an optional portion to this study, we will examine whether allergy skin testing can predict whether someone will develop a hypersensitivity reaction.

Participants who develop a moderate to severe allergic reaction to oxaliplatin will be invited to participate in an additional portion of the study examining a desensitization process. This part of the study will examine whether a desensitization process can prevent future hypersensitivity reactions to oxaliplatin in patients who previously developed moderate to severe hypersensitivity reactions and allow therapy with oxaliplatin to continue.

DETAILED DESCRIPTION:
* Participants will come in for chemotherapy treatment as scheduled by their oncologist. The frequency of the visits will depend upon the chemotherapy regimen the participant is receiving.
* With each visit, the participants will have a physical exam and will be asked questions about their general health and specific questions about any problems that they might be having and any medications they may be taking. At each of these visits, routine blood work will be taken to monitor the participant's health.
* While the participants are receiving oxaliplatin, the infusion nurse will monitor them for any evidence of hypersensitivity reaction. Participants will also leave with a diary to record any symptoms that may occur for 24 hours after they have completed the infusion of oxaliplatin.
* In the optional portion of the study, participants will undergo allergy skin testing in the Allergy Service at Brigham and Women's Hospital The skin testing will be done at three time points: before the first dose of oxaliplatin, before the 5th dose of oxaliplatin, and before the 10th dose of oxaliplatin.
* Desensitization is a method used to help a person with an allergy tolerate exposure to a specific allergic agent. Desensitization to a medication such as oxaliplatin involves giving the medication in slowly increasing amounts, starting with tiny doses, and ending with the full dose prescribed by the physician. Patients participating in this part of the study will have the desensitization at Brigham and Women's Hospital in the Medical Intensive Care Unit (ICU or MICU) to ensure close supervision. Desensitization to oxaliplatin involves a multi-step procedure where the oxaliplatin dose is started at very small doses and the rate of infusion is increased every 15 minutes until the "target rate" is achieved. This rate is then maintained until the full dose of medication has been infused. This usually takes approximately 6 hours if no adverse reactions are experienced.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically or cytologically confirmed colorectal cancer, esophageal cancer, gastric cancer, small bowel cancer, hepatobiliary cancer and pancreatic cancer
* Patients must be eligible for treatment with oxaliplatin
* ECOG Performance Status of 2 or less
* Adequate bone marrow, renal and hepatic function as outlined in the protocol
* Patients must have recovered from both the acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy
* Patients may participate in monitoring for hypersensitivity and skin testing if they are receiving oxaliplatin as part of another clinical trial and allowed by that trial. Patients cannot receive oxaliplatin through the desensitization protocol if they are part of another clinical trial.

Exclusion Criteria:

* Prior treatment with oxaliplatin
* Active infection or with a fever of 101.3 or higher within 3 days of the first scheduled days of protocol treatment
* Patients with active CNS metastases. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for greater than 3 weeks are eligible.
* Patients with known hypersensitivity to any of the components of oxaliplatin or chemotherapeutic agent used in combination with oxaliplatin
* Patients who have received radiotherapy to more than 25% of their bone marrow; or patients who received any radiotherapy within 4 weeks of study entry
* Peripheral neuropathy of grade 2 or higher
* Patients who are pregnant or lactating
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the patient's ability to sign informed consent, cooperate and participate in teh study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at Dana-Farber Cancer Institute with the chemotherapy drug oxaliplatin.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
To determine prospectively the incidence and severity of hypersensitivity reactions to oxaliplatin among patients beginning treatment with oxaliplatin during a two-year observation period. | 2 years

SECONDARY OUTCOMES:
To determine the relationship between cumulative dose of oxaliplatin and duration of therapy and development of hypersensitivity reactions. | 2 years
To determine the ability of oxaliplatin skin testing to identify patients at risk for developing hypersensitivity reactions. | 2 years
To determine the safety and efficacy of a rapid desensitization protocol to allow responding patients with moderate to severe hypersensitivity reactions to oxaliplatin to continue therapy with the drug. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Chan, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States